CLINICAL TRIAL: NCT00266591
Title: Single Center TOPAMAX� (Topiramate) Monotherapy Trial in Subjects With Refractory Partial Onset Seizures
Brief Title: A Study of the Efficacy and Safety of Topiramate Treatment in Patients With Epilepsy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR005470
Record Dates: First submitted 2005-12-16; First posted 2005-12-19 (Estimated); Last update posted 2011-06-08 (Estimated); Status verified 2011-01

CONDITIONS: Epilepsy; Seizures
Keywords: Epilepsy; Seizures; Topiramate; Prophylaxis; Antiepileptic; Epileptic seizures; Partial seizure disorder; Brain disease
MeSH Terms: conditions — Epilepsy; Seizures; Epilepsies, Partial; Brain Diseases | interventions — Topiramate

INTERVENTIONS:
Drug: topiramate

SUMMARY:
The purpose of this study is to evaluate the effectiveness and safety of topiramate (an antiepileptic medication) in patients with epilepsy.

DETAILED DESCRIPTION:
Epilepsy is a disease characterized by seizures, which are abnormal electrical discharges in the brain that temporarily disrupt normal brain function. Seizures are classified as "generalized," originating in both sides of the brain at the same time, or "partial onset," starting in one area of the brain. Antiepileptic medications, such as topiramate, are selected based on a patient's seizure type. The specific type of seizure is not always obvious at the time of diagnosis. This is a randomized, double-blind, parallel-group study to evaluate the effectiveness and safety of two doses of topiramate (100 or 1000 mg per day) in patients with partial onset seizures. The study is composed of three phases: an 8-week baseline phase during which patients take their standard antiepileptic drugs, a 1-week open-treatment phase during which patients continue standard antiepileptic drugs and add on topiramate (100 mg/day), and a double-blind treatment phase. The double-blind phase is divided into two periods: a 5-week conversion period and an 11-week treatment period with topiramate. In the conversion period, patients gradually discontinue their baseline antiepileptic drugs. Those assigned to the topiramate 1000 mg/day group start by taking the 100 mg/day dose and gradually increase to 1000 mg/day (or to their maximum tolerated dose) over a 5-week period. Patients assigned to topiramate 100 mg/day receive one 100 mg tablet (plus placebo tablets to maintain the blind during the 5 week period). Patients in both groups continue with their dose for the 11-week treatment period. Patients are provided with diaries to record information regarding any seizures occurring during the study. The primary assessment of effectiveness is the amount of time the patient receives topiramate in the double-blind treatment phase before exiting (withdrawing) from the study. Four exit criteria for withdrawal are designed to correspond to therapeutic failure and to ensure subject safety: i) a doubling of the average monthly (28-day) seizure frequency compared to baseline; ii) a doubling of the highest two-day seizure frequency that occurred during baseline; iii) a single generalized seizure if none occurred during the baseline phase; iv) or prolongation of generalized seizure duration (serial seizures or status epilepticus) as compared to the baseline phase seizure duration and requiring intervention. Safety assessments during the study include the frequency and severity of adverse events, results of clinical laboratory tests (hematology, biochemistry, and urinalysis), blood gastrin levels, measurements of vital signs and body weight, patient global evaluations of study drug tolerability, neurologic examinations, neuropsychologic tests, and physical examination findings. Based on the investigator's judgment, all patients completing the study could be enrolled into an open-label extension phase, during which patients know the identity and dose of topiramate. The study hypothesis is that the 1000 mg/day dose of topiramate is superior to the 100 mg/day dose in the amount of time before patients exit (withdraw based on pre-established exit criteria corresponding to therapeutic failure) from the double-blind phase. 100 mg/day group: one Topiramate 100 mg oral tablet (plus placebo tablets to maintain the blind) for 16 weeks. 1000 mg/day group: starting with one Topiramate 100 mg oral tablet and gradually increasing to 1000 mg/day (or maximum tolerated dose) over 5 weeks, and continuing that dose for 11 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Body weight >90 pounds
* documented history of frequent partial onset seizures
* at least four partial onset seizures per month while taking a constant antiepileptic drug dosage during the screening period
* a recent history of maintenance on 1 or 2 standard antiepileptic drugs
* females must be postmenopausal for at least 1 year, or if of childbearing age, be sexually abstinent, surgically sterile, or using adequate birth control measures, and have a negative pregnancy test before study entry.

Exclusion Criteria:

* Patients who do not have epilepsy, such as patients with treatable causes of seizure (for example, cancer or active infection)
* have a documented history (previous 3 months) of generalized status epilepticus while receiving anticonvulsant medication (status epilepticus is a prolonged seizure or seizures repeated frequently over 20 to 30 minutes so that recovery between episodes does not occur)
* have seizures occurring in only clustered patterns (numerous seizures over a short period of time)
* a significant history (within 2 years) of medical disease (heart, kidney, hormone, gynecologic, muscle, bone, gastrointestinal, metabolic, liver diseases or cancer with a metastatic potential)
* history of alcohol or drug abuse history within the past 1 year.

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 1992-10; Study Completion 1997-04 (Actual)

PRIMARY OUTCOMES:
Time to patient exit (withdrawal) from the double-blind phase of the study, based on 4 pre-established exit criteria corresponding to therapeutic failure.

SECONDARY OUTCOMES:
Investigator and patient global evaluation of the clinical response; safety evaluations conducted throughout the study (incidence and severity of adverse events, changes in physical and neurological examinations, laboratory tests)

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.

REFERENCES:
- See also: A study of the effectiveness and safety of topiramate monotherapy treatment in patients with epilepsy — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=649&filename=CR005470_CSR.pdf